CLINICAL TRIAL: NCT01731990
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study of the Safety, Tolerability and Effects on Arterial Structure and Function of ACZ885 in Patients With Intermittent Claudication.
Brief Title: Safety, Tolerability and Efficacy of ACZ885 on Leg Artery Structure in Patients With Peripheral Artery Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study got terminated based on result from primary endpoint analysis
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CACZ885M2201; 2012-001427-12
Record Dates: First submitted 2012-11-18; First posted 2012-11-22 (Estimated); Results first posted 2017-08-22 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral artery disease; Intermittent claudication; magnetic resonance imaging
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Canakinumab (ACZ885) (Experimental): Monthly subcutaneous doses of Canakinumab 150 mg/1 mL for 12 months
  Interventions: Drug: Canakinumab (ACZ885)
- Placebo (Placebo Comparator): Monthly subcutaneous doses of placebo of Canakinumab 150 mg/1 mL for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canakinumab (ACZ885) — Dosage form: solution for injection Strength: 150 mg/1 mL Mode of administration: subcutaneous use.
  Arms: Canakinumab (ACZ885)
Drug: Placebo — Matching placebo of Canakinumab
  Arms: Placebo

SUMMARY:
This study was designed to assess the safety, tolerability and efficacy of ACZ885 on the leg artery structure and physical activity in patients with atherosclerotic peripheral artery disease and leg pain from walking.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a signed informed consent form.
* Must be between the ages of 18 and 85
* Must experience leg pain associated with walking and have an ankle brachial index between 0.40 and 0.9
* Must be on stable aspirin and statin doses for at least 6 weeks
* Blood pressure within ranges specified in the protocol
* Able to communicate well with the Investigator and understand and comply with the study procedures

Key Exclusion Criteria:

* Recent use of any other experimental drugs
* Pregnant or nursing women
* Women of child bearing potential unless willing to use contraception as detailed in the protocol
* Cannot walk 15 meters (50 feet)
* People on restricted medications as listed in the protocol
* Any open or non-healing wounds with 3 months of study start or infection within 2 weeks or study start
* Significant heart disease
* Uncontrolled diabetes
* Significant kidney or liver disease
* Live vaccinations within 3 months of study start
* History of untreated tuberculosis or active tuberculosis (TB)
* Patients with metal in their body (excluded due to MRI scan) as detailed in the protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-10-30 (Actual); Primary Completion 2016-08-04 (Actual); Study Completion 2016-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (7):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Lutherville, Maryland
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Richmond, Virginia
- Germany (4):
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
- Novartis Investigative Site, Amman, Jordan

REFERENCES:
- [Derived] Russell KS, Yates DP, Kramer CM, Feller A, Mahling P, Colin L, Clough T, Wang T, LaPerna L, Patel A, Lawall H, Shennak MM, Fulmer J, Nikol S, Smith WB, Muller OJ, Ratchford EV, Basson CT. A randomized, placebo-controlled trial of canakinumab in patients with peripheral artery disease. Vasc Med. 2019 Oct;24(5):414-421. doi: 10.1177/1358863X19859072. Epub 2019 Jul 5. PMID 31277561
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=162

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 38 patients were enrolled into the study.
Period: Overall Study
Arm/Group | Canakinumab (ACZ885) | Placebo
Started | 18 ("Started" indicates Safety and Pharmacodynamics set .) | 20
Completed | 14 | 12
Not Completed | 4 | 8
Not completed — Adverse Event | 1 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol deviation | 1 | 2
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: safety analysis set: All patients that received any study drug were included in the safety analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Canakinumab (ACZ885) | Placebo | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (8.64) | 63.5 (7.98) | 64.7 (8.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Mean Vessel Wall Area Ratio of 12 Months to Baseline
Description: Peripheral artery wall area (superficial femoral artery) measured using Magnetic Resonance Imaging (MRI) cross-section slices. Mean vessel wall area (mm^2) was derived by converting total plaque volume (TPV) (mL) of the vessel to mm^3 by multiplying by 1000, dividing by the number of slices used for the volume calculation, and dividing by the thickness of a slice (3 mm). Least squares mean for ratio of 12 months to baseline was measured from repeated measures mixed effect model with visit, treatment, the treatment-by-visit interaction, baseline and the visit-by-baseline interaction as fixed effects.
Time Frame: Baseline, 12 months post-dose
Population: The pharmacodynamics (PD) analysis set included all patients with available PD data and no protocol deviations with relevant impact on PD data. Patients who underwent iliac/femoral stenting were removed from all data points that occurred after this procedure in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Canakinumab (ACZ885) | Placebo
Number analyzed (Participants) | 12 | 9
Ratio | 1.05 (0.03) | 0.99 (0.04)
Statistical Analysis 1: Comparison: Canakinumab (ACZ885) vs Placebo; Test type: Superiority or Other; p = 0.284, Mixed Models Analysis; Treatment effect for ratio to placebo = 1.06, 90% CI 2-sided [0.97 to 1.15]

2. Secondary Outcome: Number of Patients With Adverse Events in 12 Months
Description: Summary statistics on adverse event is reported. It is categorized as number of patients in total adverse events (non serious and serious AEs), serious adverse event, death.
Time Frame: Baseline to 12 months post-dose
Population: All patients that received any study drug were included in the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab (ACZ885) | Placebo
Number analyzed (Participants) | 18 | 20
Participants
  Total Adverse events | 16 | 20
  Serious Adverse events | 10 | 10
  Death | 1 | 0

3. Secondary Outcome: Serum Amyloid A (SAA) Level Ratio of 12 Months to Baseline
Description: Least squares mean for ratio of 12 months to baseline was measured from repeated measures mixed effect model with visit, treatment, treatment-by-visit interaction, baseline and the visit-by-baseline interaction as fixed effects.
Time Frame: Baseline, 12 months post-dose
Population: The PD analysis set included all patients with available PD data and no protocol deviations with relevant impact on PD data. Patients with baseline and 12 month data are included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Canakinumab (ACZ885) | Placebo
Number analyzed (Participants) | 15 | 13
Ratio | 0.62 (0.12) | 0.79 (0.17)

4. Secondary Outcome: High Sensitivity C-reactive Protein (hsCRP) Ratio of 12 Months to Baseline
Description: as for outcome 3
Time Frame: Baseline, 12 months post-dose
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Canakinumab (ACZ885) | Placebo
Number analyzed (Participants) | 15 | 13
Ratio | 0.62 (0.14) | 0.83 (0.20)

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse events are reported in this record from First Patient First Treatment until Last Patient Last Visit.
Arm/Group | Canakinumab (ACZ885) | Placebo
Serious Adverse Events (participants affected / at risk) | 10/18 | 10/20
Other Adverse Events (participants affected / at risk) | 16/18 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (ACZ885) (N=18) | Placebo (N=20)
Angina pectoris (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Mesenteric arterial occlusion (Gastrointestinal disorders) | 1 | 0
Mesenteric arteriosclerosis (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 2
Abscess limb (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary vascular disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 3 | 2
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (ACZ885) (N=18) | Placebo (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Plasma cell disorder (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 2 | 1
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 2 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Goitre (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 2 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Oesophageal mucosa erythema (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Drug intolerance (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 2
Feeling cold (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 2
Conjunctivitis viral (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 4
Otitis media (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 4
Urinary tract infection (Infections and infestations) | 1 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 0
Oesophagogastroduodenoscopy abnormal (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Areflexia (Nervous system disorders) | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0
Genital pain (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 1
Lichen nitidus (Skin and subcutaneous tissue disorders) | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin plaque (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Aortic thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
Study was terminated after the third interim analysis based on result from primary outcome analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.